CLINICAL TRIAL: NCT02411409
Title: Impact of the CommunityRx Program on Health, Service Utilization and Costs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-0771
Record Dates: First submitted 2014-07-25; First posted 2015-04-08 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Connecting Patients to Self-care Resources
Keywords: Health Information Technology (HIT); self-care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): This group of patients receives the HealtheRx.
  Interventions: Behavioral: HealtheRx
- Control group (No Intervention): This group of patients does not receive the HealtheRx

INTERVENTIONS:
Behavioral: HealtheRx — The HealtheRx is a prescription for community self-care resources. It includes a printed list of self-care resources provided to the patient at an ambulatory visit and tailored based on data from the electronic medical record.
  Arms: Intervention group

SUMMARY:
The CommunityRx system generates patient-centered e-prescriptions for community services (HealtheRx) via an interface between the electronic health records (EHR) and a comprehensive community resource database. Based on a patient's diagnoses, a HealtheRx will be printed automatically at the end of the ambulatory care visit and will provide patients with a customized map and/or list of places in their community that provide health and social services as well as contact information for a local community health worker who can provide limited case management support. The CommunityRx program aims to promote: 1) better healthcare, 2) better health, and 3) lower cost. The purpose of this research is to systematically evaluate the impact of CommunityRx on health outcomes as well as health care service utilization and total cost of care for Medicaid, Medicare and other beneficiaries. The investigators hypothesize that beneficiaries who participate in the CommunityRx intervention will experience better healthcare, better health and lower total cost of care.

ELIGIBILITY:
Inclusion Criteria:

* Intervention group eligibility: Patients receiving ambulatory care at a clinical site connected to CommunityRx who live in the CommunityRx geography. Control group eligibility: Patients receiving care at a clinical site connected to CommunityRx who live outside the CommunityRx geography.

Exclusion Criteria:

* Patients receiving care at a clinical site not connected to CommunityRx.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 113295 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Change in cost per beneficiary per year | Annual, up to 6 years
  Cost per beneficiary per year

SECONDARY OUTCOMES:
Change in emergency department visit rate | Every 3 months, up to 72 months
  Hospital emergency department visit rate, overall and for patients diagnosed with a) diabetes, b) hypertension, and c) asthma
Change in HbA1c control | Every 3 months, up to 72 months
  Percentage of patients 18-75 years of age with diabetes (type 1 or type 2) who had hemoglobin A1c > 9.0 %.
Change in controlling high blood pressure | Every 3 months, up to 72 months
  % of patients >=18 years old with hypertension diagnosis and a most recent BP measure <140/90mg
Change in body mass index | Every 3 months, up to 72 months
  Percentage of patients overweight or obese (BMI >=25.0 and <30, BMI >=30)
Change in inpatient admission rate | Every 3 months, up to 72 months
  Average number of in patient admissions per person
Change in participant satisfaction (percentage of participants reporting they are satisfied with the HealtheRx) | Every 3 months, up to 60 months
  Program participant satisfaction survey, percentage of participants reporting they are satisfied with the HealtheRx
Change in provider satisfaction ( percent of providers reporting they are satisfied with the HealtheRx system) | Every 6 months, up to 60 months
  Provider satisfaction survey, percent of providers reporting they are satisfied with the HealtheRx system
Change in rate of participant use of community-based service providers listed on HealtheRx | Every 3 months, up to 60 months
  Program participant survey, percent of participants who report using at least 1 service listed on their HealtheRx
Change in HealtheRx reach (proportion of the population in the geography who receive at least 1 HealtheRx) | Every 3 months, up to 60 months
  The proportion of the population in the geography who receive at least 1 HealtheRx
Change in HealtheRx delivery (providers communicate to patients about the HealtheRx) | Every 3 months, up to 60 months
  providers communicate to patients about the HealtheRx
Change in HealtheRx usefulness (participant survey, the percent of program participants who report that their HealtheRx is useful) | Every 3 months, up to 60 months
  Program participant survey, the percent of program participants who report that their HealtheRx is useful
Change in HealtheRx Understandability (participant survey, the percent of program participants who report that their HealtheRx is easy to understand) | Every 3 months, up to 60 months
  Program participant survey, the percent of program participants who report that their HealtheRx is easy to understand
Change in information sharing (participant survey, the percent of program participants who report that they shared information about the HealtheRx with someone else) | Every 3 months, up to 60 months
  Program participant survey, the percent of program participants who report that they shared information about the HealtheRx with someone else
Change in knowledge about resources (participant survey, the percent of program participants who report that they did not know about some of the places listed on their HealtheRx) | Every 3 months, up to 60 months
  Program participant survey, the percent of program participants who report that they did not know about some of the places listed on their HealtheRx
Change in provider confidence in serving social needs (Provider satisfaction survey,) | Every 6 months, up to 60 months
  Provider satisfaction survey, the proportion of providers reporting they are confident in their ability to serve their patients social needs

OTHER OUTCOMES:
Change in technical problems with the CommunityRx system (e.g., number of times system does not work properly) | Every 3 months, up to 60 months
  The number of technical problems experienced with the CommunityRx system (e.g., number of times system does not work properly)
Change in % of eligible patients receiving a HealtheRx | Every 3 months, up to 60 months
  CommunityRx database and electronic medical records, the proportion of eligible patients who receive a HealtheRx
Change in number of places mapped (community organizations, identified in the geographic region) | Every year, up to 6 years
  Number of places, or community organizations, identified in the geographic region
Change in number of CommunityRx reports delivered (Number of CommunityRx reports created and given to community organizations) | Every 3 months, up to 60 months
  Number of CommunityRx reports created and given to community organizations
Change in number of times a community health information specialist is contacted (CHIS call tracker) | Every 3 months, up to 60 months
  CHIS call tracker, number of times a program participant contacted a CHIS
Change in referrals by service type (number of referrals, or number of times a service was listed on a HealtheRx) | Every 3 months, up to 60 months
  CommunityRx database, number of referrals, or number of times a service was listed on a HealtheRx
Change in services identified (number of services identified as available at community organizations0 | Every 3 months, up to 60 months
  Service level survey, count of number of services identified as available at community organizations

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Lindau, MD, MAPP, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States